CLINICAL TRIAL: NCT07383129
Title: Early Brochoscopic Intervention Versus Conventional Management in the Treatment of Acute Lung Collapse Among Critically Ill Children in the Pediatric Intensive Care Unit
Brief Title: Brochoscopic Intervention Versus Conventional Management in Acute Lung Collapse in the Pediatric Intensive Care Unit
Acronym: picu
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Samy, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-462-2025; MD-462-2025 (Other: cair0 university faculty of medicine- research ethics committee.)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Bronchoscopes; Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early broncoscopic intervention (Experimental): patients with acute lung collapse receive Patients with acute lung collapse receive early flexible bronchoscopy in addition to standard pediatric intensive care management.
  Interventions: Procedure: bronchoscope
- conventional management (Active Comparator): patients with acute lung collapse receive Patients with acute lung collapse receive conventional intensive care unit protocol without early broncoscopy
  Interventions: Other: chest physiotherapy and suction

INTERVENTIONS:
Procedure: bronchoscope — This RCT stands out by randomizing refractory pediatric atelectasis (post-48h failed recruitment) to fiberoptic bronchoscopy with active inflation vs. optimized conventional care (suctioning, physiotherapy ± cough assist) with crossover.
  Unique Aspects: Targets true refractory cases after standardized recruitment, unlike diagnostic FFB series (mucus plugs ~50%) or elective bronchoscopy. Uses flexible scope for therapeutic inflation, not rigid removal, CPAP-endobrochial in CHD, dornase instillation, or unstructured physio alone.
  Differentiation: 5-day pulmonologist-assessed radiographic/clinical endpoint tests superiority absent in pediatric RCTs; powers ventilation-free days/VAP. Isolates bronchoscopy in mixed PICU etiologies. (578 chars)
  Arms: early broncoscopic intervention
Other: chest physiotherapy and suction — Conventional Management Endotracheal suctioning, chest physiotherapy (percussion/postural drainage), ± cough assist device (positive/negative pressure cycles). recruitment maneuvers; assessed day 5 for clinical/radiographic response.
  Arms: conventional management

SUMMARY:
This prospective RCT at Cairo University Children Hospitals enrolls critically ill pediatric patients (intubated, NIV, or post-extubation) with lung atelectasis unresponsive to 48 hours of conventional recruitment. Randomization uses computer-generated sealed envelopes: Group A receives bronchoscopy with active inflation; Group B gets suctioning, chest physiotherapy ± cough assist. Crossover permitted after 5 days failure or if unsafe; pulmonologist assesses. Data covers personal history (age, sex, weight, residency) and clinical details (PICU diagnosis, symptoms/duration).

Strengths include bias-minimizing allocation, ethical flexibility, and standardized baselines. Suggested expansions: ventilation parameters (mode, FiO2, PEEP), atelectasis scoring (X-ray/US), outcomes (P/F ratio, LOS, VAP), and safety metrics for power (targeting 20-30% non-response) to align with PALICC-2. (612 chars)

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial (RCT) enrolling critically ill patients intubated , on non-invasive ventilation or post-extubation with lung atelectasis admitted at pediatrics emergency and intensive care units, Cairo University Children Hospitals, identified by treating medical team.

Patient randomization will be done by a computer-based generation and serial sealed enveloped numbers was taken for the patients. Assessment will be done by a pediatric pulmonologist. All patients will be subjected to routine initial conventional lung inflation and recruitment maneuvers.

For those non inflatable lungs within 48 hours of conservative measures, they will be divided into two groups, group A: patients will undergo bronchoscopic intervention and active lung inflation, and group B: managed using conventional therapies, suctioning, chest physiotherapy, with or without the aid of a cough assisted device , in case of no clinical or radiological improvement after 5 days this is considered failure of conventional methods patients in this group may take a chance to do bronchoscopy (Oh's Intensive Care Manual, 9th ed., 2023).

Whenever the randomly assigned therapy is considered to be failed or unsafe to be continued, the treating physician will discontinue the randomization and continue with the appropriate treatment modality according to the patients need.

ELIGIBILITY:
Inclusion Criteria:

* Radiological evidence of partial or complete lung collapse (PICU admission or during stay).

Intubated, on non-invasive ventilation, or high velocity oxygen.

Exclusion Criteria:

* obstructive collapse from endobronchial foreign body or tissue. Extrabronchial compression (tumor, lymphadenopathy, pleural effusion/pneumothorax).

Bronchoscopy contraindications: severe refractory hypoxemia, hemodynamic instability, uncorrected coagulopathy.

Musculoskeletal causes (e.g., scoliosis) or congenital lung diseases (e.g., lobar emphysema).

Ages: 1 Month to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of radiological lung re-expansion at day 5. | 12 month
  Assessed t via chest X-ray comparison (pre/post-intervention), defining success as ≥50% reduction in atelectasis opacity/area for partial collapse or full re-aeration for complete collapse. Captures therapeutic efficacy post-bronchoscopy (Group A immediate) vs. conventional care (Group B day 5), aligning with trial power on LOS reduction. (312 chars)

CONTACTS AND LOCATIONS:
Overall Officials: fatma samy, masters, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt